CLINICAL TRIAL: NCT04929522
Title: Success Rate of 4 Injection Protocols for Mandibular First Molars With Symptomatic Irreversible Pulpitis: A CONSORT Randomized Triple-blind Clinical Trial
Brief Title: Success Rate of 4 Injection Protocols for Mandibular First Molars With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shehab El Din Mohamed Saber, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-REC IM061101
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Root Canal Infection
Keywords: intra-osseous injection; PDL injection; IANB
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: This study was a prospective, randomized, parallel, triple blinded, clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation concealment mechanism: The sequentially generated numbers were placed in opaque envelopes until the intervention was conducted, and each participant was asked to select an envelope that determines which group of intervention was assumed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IANB/inferior alveolar nerve block (Active Comparator): patients will be given standard IANB with 3.6 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  Interventions: Procedure: local anesthesia
- IANB+IO (Active Comparator): patients will be given standard IANB plus an intra-osseous with 3.6 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  Interventions: Procedure: local anesthesia
- IANB+PDL (Active Comparator): patients will be given standard IANB plus a PDL injection with 3.6 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  Interventions: Procedure: local anesthesia
- IANB+BI (Active Comparator): patients will be given standard IANB plus a BI injection with 3.6 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  Interventions: Procedure: local anesthesia

INTERVENTIONS:
Procedure: local anesthesia — technique for local anesthesia

SUMMARY:
Achieving profound anesthesia during endodontic treatment of mandibular molars with symptomatic irreversible pulpitis is still a demanding clinical challenge. therefore, the success Rate of 4 Injection protocols for Mandibular First Molars with Symptomatic Irreversible Pulpitis was evaluated clinically in a randomized triple-blind trial

DETAILED DESCRIPTION:
Trial design This study was a prospective, randomized, parallel, triple blinded, clinical trial. The present trial design methodology conforms to the CONSORT guidelines for reporting randomized clinical trials.Participants A sample size calculation was performed based on the study by (Kanaa M, Whitworth JM, Meechan JG. A Prospective Randomized Trial of Different Supplementary Local Anesthetic Techniques after Failure of Inferior Alveolar Nerve Block in Patients with Irreversible Pulpitis in Mandibular Teeth. J Endod 2012;38:421-425). This research was based on a type I error of 0.05 and a power of 0.8 and indicated that ideally a sample size of 36 in each group would be required to detect a 20% difference in the success rate of the test groups. To increase the validity of the study, 40 subjects in each group were considered.Ethical considerations This trial was conducted with the approval of the institutional review of board (IRB) of the ethics committee at the Faculty of Dentistry, Ain Shams University, Cairo, Egypt (FDASU-REC 772019). Patients signed a printed informed consent form after explanation of the treatment procedure and associated possible adverse effects of the proposed interventions such as discomfort, pain, anesthetic failure and systemic side effects at this stage. Randomization To ensure random selection, participants were allocated randomly into four groups with1:1 allocation ratio by using computer generated randomization (www.randome.org). The sequence was therefore generated.

Allocation concealment mechanism: The sequentially generated numbers were placed in opaque envelopes until the intervention was conducted, and each participant was asked to select an envelope that determines which group of intervention was assumed.

Implementation: Co-researcher used computer generated randomization for participants who achieve eligibility criteria and accordingly participants were enrolled in either of the groups under study.

Blinding Both the participants, the operator who initiated endodontic treatment and monitored the pain, and the statistician were blinded to the anesthetic techniques used.

Intervention Diagnosis was confirmed through history reporting spontaneous pain, a moderate to severe painful response that persists after thermal stimulation, a prolonged response to cold testing with Endo-Ice (1,1,1,2 tetrafluoroethane; Hygenic Corp, Akron, OH), absence of percussion sensitivity and the periapical aspect of the tooth in the bidimensional periapical radiograph was normal. Matching vital contralateral teeth were also tested to ensure an accurate diagnosis and to serve as controls. To prevent bias, this diagnostic step was performed by one investigator (AH), while another investigator (DK) was responsible for administration of all anesthetic injections (DK), and a third investigator (SS) was responsible for root canal treatment procedures and pain recording. All investigators have a minimum of 12 years of clinical experience in endodontics.

One hundred and eighty-five patients consecutively visited were assessed for eligibility. Twenty-five patients were excluded for different reasons and the others (eighty-four female and seventy-six male patients) were allocated to the trial (Figure 1) and randomly assigned into 4 groups (n=40) as follows:

Group 1 (IANB): After determining the injection site and aspiration, 3.6ml of the anesthetic solution was administered using the standard inferior alveolar nerve block (IANB), this was considered the control group.

Group 2 (IANB + IO): A standard IANB was administered the same as for Group 1, followed by a supplemental intraosseous infusion (IO) injection using the Anesto system (W&H Dentalwerk Bürmoos, Austria). To ensure comfort during the procedure, 0.1ml of anesthetic solution was infiltrated at the perforation site using the standard syringe. The perforation site was selected near the junction of the attached and unattached gingival tissues, immediately distal to the first molar. Perforation was accomplished by operating the Anesto handpiece at full speed, with constant moderate pressure maintained until the perforator was felt to 'drop' into the cancellous bone. 1.8mL of the anesthetic solution was then deposited over a 60-second period. The Anesto handpiece was again retracted and, with the perforator rotating, removed from the injection site.

Group 3 (IANB + PDL): A standard IANB was administered the same as for groups 1 and 3, followed by a supplemental periodontal ligament (PDL) injection. The needle was wedged with force into the PDL space between the tooth and the alveolar crest of the bone, at 30-degrees to the long axis of the tooth. The thumb and index fingers of the left hand supported the needle to prevent buckling. The handle of the syringe was squeezed firmly until backpressure was achieved. Then a total of 1.8ml of the anesthetic solution were injected mesially and distally to the treated molar.

Group 4 (IANB + BI): A standard IANB was administered the same as for groups 1, 2 and 3, followed by a supplemental buccal infiltration at the buccal side of the affected tooth. A total of 1.8ml of the anesthetic solution were injected halfway the mesiodistal width of the clinical crown.

IANB, PDL and BI injections were performed with a conventional dental syringe (indicate the brand) and a 27-G needle at a rate of 2 mL/min. The anesthetic solution used for all techniques was Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain). The efficacy of anesthesia was determined by the following: (1) confirmation of lip numbness, (2) negative response to Endo-Ice, (3) negative response to the maximum output of the electric pulp tester (Parkell, Edgewood, NY, USA).

Root canal treatment procedure was later initiated, and the patients were asked to rate their pain using a visual analogue scale (VAS). Pain was scored as follows: Score 0, no pain; Score 1, mild pain; Score 2, moderate pain; or Score 3, severe pain. After rubber dam placement and during caries removal, access preparation and pulpectomy, success of the anesthetic technique was determined by VAS. The technique was considered as a 'success' when the patient reported no pain (VAS = 0 or 1) and as a 'failure' otherwise (VAS >1).

Heart rate changes were monitored with a finger pulse oximeter (Medlinket, Shenzhen Med-link Electronics, Shenzhen, China). It was recorded from 2 min before to 5 min after injection, at 30-s intervals. The mean heart rate for each injection was recorded.

Statistical analysis All analyses were undertaken with IBM SPSS Statistics (SPSS 26.0; SPSS Inc., Chicago, IL). The anesthetic success rates were analyzed using the chi-square test. Age differences were analyzed using One Way ANOVA, gender differences were analyzed using the Fischer Exact test while heart rate changes were analysed with Kruskal Wallis test, being non-normally distributed. Statistically significant differences were set at the P < 0.05 level

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study were healthy males and females
* (Category: American Society of Anesthesiologists class 1)
* aged 21-49 years
* with no physical disability, facial paresthesia or psychological problems
* presenting with a single vital mature mandibular first molar, with signs and/or symptoms of symptomatic irreversible pulpitis

Exclusion Criteria:

* Pregnant women
* patients who took analgesics or other medications that would alter the inflammatory response of the pulp or provide analgesia 6- hours pre-operatively
* those with known sensitivity to the pharmaceuticals used in this trial.
* those with pathological periodontal pockets

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel Rahman Hashem, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IANB/Inferior Alveolar Nerve Block | IANB+IO | IANB+PDL | IANB+BI
Started | 40 | 40 | 40 | 40
Completed | 40 | 40 | 40 | 40
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IANB/Inferior Alveolar Nerve Block: patients were given a standard IANB with 3.6 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
- IANB+IO: patients were given a standard IANB (1.8 ml) followed by an intra-osseous supplemental injection (1.8 ml) Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
- IANB+PDL: patients were given a standard IANB (1.8 ml) followed by a PDL supplemental injection (1.8 ml) with Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
- IANB+BI: patients were given a standard IANB (1.8 ml) followed by a Buccal infiltration injection (1.8 ml) with Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
- Total: Total of all reporting groups
Arm/Group | IANB/Inferior Alveolar Nerve Block | IANB+IO | IANB+PDL | IANB+BI | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 40 | 40 | 160
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 26 | 23 | 102
  Male | 15 | 12 | 14 | 17 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 40 | 40 | 40 | 40 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Injection Technique Assessed by Verbal Rating Scale (VRS)
Description: the patients were asked to rate their pain using a Verbal rating scale (VRS). Pain was scored as follows: Score 0, no pain; Score 1, mild pain; Score 2, moderate pain; or Score 3, severe pain. After rubber dam placement and during caries removal, access preparation and pulpectomy, success of the anesthetic technique was determined by NRS. The technique was considered as a 'success' when the patient reported no pain (VRS = 0 or 1) and as a 'failure' otherwise (vRS >1).
Time Frame: 15 minutes from delivery of anesthesia
Measure: Count of Participants; unit: Participants
Groups:
- IANB+IO: patients were given a standard IANB (1.8 ml) followed by an intra-osseous injection with 1.8 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
- IANB+PDL: patients were given standard IANB (1.8 ml) followed by a PDL injection with 1.8 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
- IANB+BI: patients were given a standard IANB )1.8 ml) followed a Buccal Infiltration injection with 1.8 ml Articaine HCL 4% with 1:100,000 adrenaline (Artinibsa, Inibsa, Barcelona, Spain).
  local anesthesia: technique for local anesthesia
Arm/Group | IANB/Inferior Alveolar Nerve Block | IANB+IO | IANB+PDL | IANB+BI
Number analyzed (Participants) | 40 | 40 | 40 | 40
Participants | 16 | 37 | 29 | 26

2. Secondary Outcome: Changes in the Heart Rate Before, During and After the Injection
Description: beat per minute measured by a finger pulse oximeter
Time Frame: assessed from 2 min before to 5 min after injection (at 30-s intervals)
Measure: Mean (Standard Deviation); unit: beat per minutes
Arm/Group | IANB/Inferior Alveolar Nerve Block | IANB+IO | IANB+PDL | IANB+BI
Number analyzed (Participants) | 40 | 40 | 40 | 40
beat per minutes
  -2 minutes | 72 (4) | 72 (5) | 71 (4) | 71 (5)
  -1.5 minutes | 71 (4) | 72 (5) | 70 (4) | 69 (4)
  -1 minute | 71 (5) | 71 (4) | 71 (5) | 70 (4)
  -0.5 minute | 72 (5) | 72 (5) | 72 (4) | 71 (3)
  0 minutes | 75 (6) | 80 (7) | 74 (5) | 72 (5)
  0.5 minute | 76 (4) | 85 (5) | 75 (6) | 72 (4)
  1 minute | 74 (5) | 84 (6) | 73 (4) | 71 (4)
  1.5 minutes | 74 (5) | 83 (7) | 73 (5) | 71 (4)
  2 minutes | 72 (4) | 80 (6) | 72 (5) | 71 (4)
  2.5 minutes | 72 (4) | 77 (5) | 72 (3) | 70 (4)
  3 minutes | 71 (3) | 74 (4) | 72 (4) | 71 (2)
  3.5 minutes | 72 (3) | 72 (4) | 72 (4) | 71 (3)
  4 minutes | 72 (4) | 71 (3) | 71 (3) | 72 (3)
  4.5 minutes | 71 (4) | 72 (3) | 71 (3) | 71 (2)
  5 minutes | 71 (3) | 71 (2) | 71 (1) | 72 (3)

ADVERSE EVENTS:
Time Frame: from 2 min before to 5 min after injection, at 30-s intervals.
Description: Only healthy individuals participated in the trial, so they were not liable to any adverse effect associated with the standard dental injections.
  Even no one complained from prolonged lip numbness.
Arm/Group | IANB/Inferior Alveolar Nerve Block | IANB+IO | IANB+PDL | IANB+BI
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT04929522/Prot_SAP_000.pdf